CLINICAL TRIAL: NCT06429930
Title: A Phase 1, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of L608 for Inhalation in Healthy Participants
Brief Title: Safety, Tolerability and Pharmacokinetics Study of L608 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmosa Biopharm Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PBI-L608-B12
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases; Pharmaceutical Solutions
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, double-blinded, single ascending dose escalation
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded, single ascending dose escalation design. After confirmation of eligibility, subjects will be randomized at a ratio of 1:1 (for sentinel dosing) followed by 5:1 for rest of the cohorts to receive the assigned dose of L608 or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L608 Liposomal inhalation suspension (Experimental): Eight participants will be enrolled in each cohort and be randomized to receive assigned dose of L608 or placebo (6:2).
  Interventions: Drug: L608 Liposomal inhalation suspension
- Placebo (Placebo Comparator): Eight participants will be enrolled in each cohort and be randomized to receive assigned dose of L608 or placebo (6:2).
  Interventions: Drug: Placebo Solution

INTERVENTIONS:
Drug: L608 Liposomal inhalation suspension — Participants will be randomized at a ratio of 1:1 (for sentinel dosing) followed by 5:1 for the rest of the cohort to receive the assigned dose of L608 or placebo.
  Arms: L608 Liposomal inhalation suspension
Drug: Placebo Solution — Participants will be randomized at a ratio of 1:1 (for sentinel dosing) followed by 5:1 for the rest of the cohort to receive the assigned dose of L608 or placebo.
  Arms: Placebo

SUMMARY:
This is the second single ascending dose study of L608 in healthy participants and is being conducted to evaluate the safety of L608 with dose level ranging from 15 μg to 30 μg.

DETAILED DESCRIPTION:
L608 inhalation Suspension (L608) is developed by Pharmosa Biopharm Inc. (PBI) as a new liposomal Iloprost formulation for inhalation use in the treatment of patients with WHO Group 1 PAH. As a liposomal formulation of iloprost, L608 is intended to reduce the dosing frequency, as well as provide sustained and selective release along with achieving therapeutically relevant iloprost level. Meanwhile, L608 is expected to mitigate burst release related local irritation and systemic side effects (e.g., hypotension due to plasma peak) in clinical practice.

This Phase I, randomized, double-blinded, placebo-controlled study will be conducted in healthy participants in New Zealand to evaluate the safety, tolerability, and pharmacokinetic of L608. The dose escalation design is applied in this study. The sentinel dosing design will be applied for all cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women aged between 18 and 65 (inclusive) at the time of Screening visit.
2. Participants with Body Mass Index (BMI) of ≥18.5 and ≤32.0 kg/m2 and weight of at least 50 kg at Screening.
3. Non-smokers or former smokers who have smoked ≤ 100 cigarettes in their lifetime and have not consumed any tobacco or tobacco-containing products for at least 3 months prior to Screening.
4. Females must not be pregnant or lactating and must use acceptable, highly effective double contraception from Screening until 3 months after the last dose of the Investigational product.

Key Exclusion Criteria:

1. Participants with contraindications or sensitivity to any components of the study treatment.
2. Participants with histories or active conditions of unexplained bleeding events, hemoptysis, abnormal bleeding tendencies, and/or coagulation disorders.
3. Participants with histories or active conditions of asthma, sleep apnea, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, bronchiectasis, bronchospasm, and/or reactive airway. Subjects who have had childhood asthma which have resolved as deemed by the PI can be considered.
4. Participants with histories or active conditions of myocardial infarction (MI), cerebrovascular accident (CVA), coronary artery disease (CAD), unstable angina, heart failure, significant cardiac arrhythmias, congenital or acquired valvular heart disease with clinically insignificant symptom, suspected lung congestion, and/or pulmonary arterial hypertension (PAH) causing by venous thromboembolism.
5. Participants with systolic blood pressure < 90 mmHg or > 140 mmHg and/or diastolic blood pressure < 50 mmHg or > 95 mmHg at Screening or check-in visit.
6. Participants with FEV1 less than 80% predicted, FVC ˂ 80% predicted, or resting oxygen saturation less than 95% at Screening or check-in visit.
7. Participants with histories of drug or alcohol abuse within 1 year prior to subject check-in (Day -1). Regular alcohol consumption defined as > 14 standard drinks per week for female and > 21 standard drinks per week for male.
8. Consumption of products containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing and products containing grapefruit and/or pomelo (shown to inhibit cytochrome P450 [CYP] 3A4 activity) within 10 days prior to drug administration, and/or participants unwilling to refrain from consumption of alcohol from 48 hours before dosing to Day 14.
9. Receipt of blood products within 2 months prior to dosing.
10. Positive results of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), and pregnancy test.
11. Blood donation or significant blood loss (>480 ml) within 3 months prior to Screening.
12. Participants unwilling to refrain from strenuous exercises from 7 days prior to dosing until the EOS visit.
13. Participants planning to receive a tattoo, body piercing, or undergo any invasive procedure during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with DLT | 7 days after administration
  DLT: Dose-limiting toxicity
Percentage of participants with TEAEs and SAEs | 2 weeks after administration
  TEAEs: treatment emergent adverse events; SAEs: serious adverse events
Frequency and severity of TEAEs and SAEs | 2 weeks after administration
  TEAEs: treatment emergent adverse events; SAEs: serious adverse events

SECONDARY OUTCOMES:
AUC0-t | 24 hours after administration
  Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration
AUC0-inf | 24 hours after administration
  Area under the plasma concentration-time curve from time 0 to infinity
%AUCextrap | 24 hours after administration
  AUC extrapolated from the last measurable concentration to infinity as a percentage of total AUC
Cmax | 24 hours after administration
  Maximum observed plasma concentration
Tmax | 24 hours after administration
  Time to reach the maximum observed plasma concentration
T1/2 | 24 hours after administration
  Apparent plasma terminal elimination half-life
CL/F | 24 hours after administration
  Apparent total plasma clearance
Vz/F | 24 hours after administration
  Apparent volume of distribution during the terminal phase
λz | 24 hours after administration
  Terminal elimination rate constant
Cmax/D | 24 hours after administration
  Dose-normalized Cmax.
AUC0-t/D | 24 hours after administration
  Dose-normalized AUC0-t.
AUC0-inf/D | 24 hours after administration
  Dose-normalized AUC0-inf.

CONTACTS AND LOCATIONS:
Locations (1):
- NZCR Ltd (New Zealand Clinical Research), Christchurch, New Zealand